CLINICAL TRIAL: NCT04150224
Title: An Open-label, Prospective Study of Safety, Tolerability, Pharmacokinetics and Food Effects of PBTZ169, 80 mg Capsules, When Used in Ascending Doses in Healthy Volunteers
Brief Title: Safety, Tolerability, Pharmacokinetics and Food Effects Study of PBTZ169
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nearmedic Plus LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: PBTZ169-Z00-C01-3
Record Dates: First submitted 2019-10-18; First posted 2019-11-04 (Actual); Results first posted 2020-02-28 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Healthy Subjects
Keywords: PBTZ169; Macozinone; Antimycobacterial; Tuberculosis; Drug Resistant Tubercolosis; MDR-TB; XDR-TB
MeSH Terms: conditions — Tuberculosis; Tuberculosis, Multidrug-Resistant; Extensively Drug-Resistant Tuberculosis | interventions — macozinone; BID protein, human

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Cohort 1 (C1A), PBTZ169 (Experimental): Two doses of PBTZ169: 640 mg OD fasted and 640 mg OD after meal. Wash-out period ≥6 days.
  Interventions: Drug: PBTZ169 640 mg OD
- Cohort 1 (C1B), PBTZ169 (Experimental): Two doses of PBTZ169: 640 mg OD after meal and 640 OD mg fasted. Wash-out period ≥6 days.
  Interventions: Drug: PBTZ169 640 mg OD
- Cohort 2 (C2), PBTZ169 (Experimental): Single dose of PBTZ169: 960 mg fasted
  Interventions: Drug: PBTZ169 960 mg SD
- Cohort 3 (C3), PBTZ169 (Experimental): Two doses of PBTZ169: 640 mg twice a day (fasted) with a 12-hour interval; total daily dose - 1280 mg
  Interventions: Drug: PBTZ169 640 mg BiD
- Cohort 4 (C4), PBTZ169 (Experimental): Single dose of PBTZ169: 1280 mg fasted
  Interventions: Drug: PBTZ169 1280 mg SD
- Cohort 5 (C5), PBTZ169 (Experimental): Multiple administration of PBTZ169: 1280 mg once a day after meal for 14 days
  Interventions: Drug: PBTZ169 1280 mg MD

INTERVENTIONS:
Drug: PBTZ169 640 mg OD — Two administrations once a day with a wash-out period: food effect
  Other Names: Macozinone (PBTZ169)
  Arms: Cohort 1 (C1A), PBTZ169; Cohort 1 (C1B), PBTZ169
Drug: PBTZ169 640 mg BiD — Twice a day fasted; 1 day of administration
  Other Names: Macozinone (PBTZ169)
  Arms: Cohort 3 (C3), PBTZ169
Drug: PBTZ169 960 mg SD — Once a day fasted
  Other Names: Macozinone (PBTZ169)
  Arms: Cohort 2 (C2), PBTZ169
Drug: PBTZ169 1280 mg SD — Once a day fasted
  Other Names: Macozinone (PBTZ169)
  Arms: Cohort 4 (C4), PBTZ169
Drug: PBTZ169 1280 mg MD — Once a day after meal, 14 doses
  Other Names: Macozinone (PBTZ169)
  Arms: Cohort 5 (C5), PBTZ169

SUMMARY:
Open-label prospective non-comparative ascending dose randomized cohort study of single and multiple oral administration of PBTZ169 (capsules 80 mg) in healthy volunteers

DETAILED DESCRIPTION:
Open-label prospective non-comparativerandomized cohort study of safety, tolerability, pharmacokinetics and the effect of food of PBTZ169 in adult healthy volunteers after single and multiple oral administration. Study was conducted in one study center in the Russian Federation. The study included two stages:

Stage 1 - single or double oral administration with dose escalation (fasted/after meal) in 5 cohorts 10 healthy volunteers each plus 5 back-up volunteers;

Stage 2 - multiple oral administration once a day after meal for 14 days in 1 cohort of 10 healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent from the volunteer.
2. Men and women aged 18-45 years, inclusive.
3. Body mass index of 18.5-30 kg/m2.
4. Verified "healthy" diagnosis based on physical examination, vital signs, standard laboratory tests (complete blood count and biochemical blood test, urine analysis) and instrumental tests (ECG, fluorography examination or X-ray examination).
5. Negative results of tests for human immunodeficiency virus (HIV), syphilis, hepatitis B (Hbs Ag) and hepatitis C (antibodies to HCV).
6. Ability to comply with all the requirements of the protocol in the opinion of the investigator.
7. Consent of the participant and his/her partner to use reliable contraceptive methods during the study and within 90 days after the end of their participation. A reliable method of contraception is a combination of a male condom with at least one of the following methods:

   * hormonal contraceptives used by the male's partner (only if she does not participate in this clinical study);
   * use of aerosols, creams, suppositories and other agents containing spermicides;
   * use of intrauterine device by female partner.

Exclusion Criteria:

1. History of allergies, including at least one episode of allergy to medications.
2. Chronic diseases of the cardiovascular, bronchopulmonary, neuroendocrine systems, ENT, as well as diseases of the gastrointestinal tract, liver, kidneys, blood, skin.
3. Hypolactasia (lactose intolerance, lactase deficiency) or glucose-galatose malabsorption in medical history.
4. Chronic eye diseases except for myopia, hypermetropia and astigmatism of mild and moderate severity.
5. Surgeries on the gastrointestinal tract (except for appendectomy done more than 1 year before screening).
6. Regular administration or use (including externally) of hormonal agent for more than 1 week less than 45 days before screening
7. Regular administration of medicinal products less than 4 weeks before screening.
8. Use of medicinal products that have a pronounced effect on liver function or hemodynamics (barbiturates, omeprazole, cimetidine, etc.) less than 30 days before screening.
9. Positive test for narcotics and psychotropic products.
10. Blood pressure after resting in supine position for at least 5 minutes above 130 mm Hg (systolic blood pressure) and 90 mm Hg (diastolic blood pressure) or below 110 mm Hg (systolic blood pressure) and 60 mm Hg (diastolic blood pressure).
11. Heart rate (according to ECG) after resting in supine position for at least 5 minutes above 90 bpm or below 60 bpm.
12. Blood donation (450 mL of blood or plasma and more) less than 3 months before the screening.
13. Acute infectious diseases less than 4 weeks before screening.
14. Administration of more than 10 units of alcohol per week (1 unit of alcohol is equivalent to 500 mL of beer, 200 mL of wine or 50 mL of a spirit) or history of alcoholism, drug abuse, substance abuse.
15. Mental diseases.
16. Smoking for three months before screening.
17. Participation in any clinical study less than 3 months before screening.
18. Planned conception or sperm donation during the study after the administration of the investigational product or within 3 months after the last administration of the product.
19. Positive pregnancy test for women.
20. Breastfeeding period.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-07-03 (Actual); Primary Completion 2018-11-23 (Actual); Study Completion 2019-02-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical hospital at the Yaroslavl station of the Open Joint Stock Company Russian Railways, Yaroslavl, Russia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Period 1: Single or double dosing (Cohorts 1-4) Period 2: Multiple dosing (Cohort 5)
Period: Overall Study
Arm/Group | Cohort 1 (C1A), PBTZ169 | Cohort 1 (C1B), PBTZ169 | Cohort 2 (C2), PBTZ169 | Cohort 3 (C3), PBTZ169 | Cohort 4 (C4), PBTZ169 | Cohort 5 (C5), PBTZ169
Started | 10 (10 healthy volunteers receiving PBTZ169 + 1 backup volunteer) | 10 (10 healthy volunteers receiving PBTZ169 + 1 backup volunteer) | 10 (10 healthy volunteers receiving PBTZ169 + 1 backup volunteer) | 10 (10 healthy volunteers receiving PBTZ169 + 1 backup volunteer) | 10 (10 healthy volunteers receiving PBTZ169 + 1 backup volunteer) | 10 (Period 2: Multple Dosing)
Completed | 10 | 10 | 10 | 10 | 10 | 10 (Period 2: Multple Dosing)
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (C1A), PBTZ169 | Cohort 1 (C1B), PBTZ169 | Cohort 2 (C2), PBTZ169 | Cohort 3 (C3), PBTZ169 | Cohort 4 (C4), PBTZ169 | Cohort 5 (C5), PBTZ169 | Total
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 10 | 10 | 10 | 10 | 60
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.2 (5.25) | 23.0 (2.26) | 23.7 (3.95) | 27.1 (5.09) | 30.1 (9.10) | 26.7 (5.01) | 26.3 (5.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 9 | 5 | 4 | 6 | 32
  Male | 5 | 7 | 1 | 5 | 6 | 4 | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 10 | 10 | 10 | 10 | 10 | 10 | 60
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 00 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events
Description: Safety and tolerability: number of (S)AEs
Time Frame: Up to last visit time point: C2, C3, C4 up to Day 7; C1 up to Day 13; C5 up to Day 21 after first drug intake
Population: Safety population
Measure: Number; unit: AEs
Groups:
- Cohort 1 (C1A+C1B), PBTZ169: Two doses of PBTZ169: 640 mg OD fasted/after meal and 640 mg OD after meal/fasted. Wash-out period ≥6 days.
  PBTZ169 640 mg OD: Two administrations once a day with a wash-out period: food effect
Arm/Group | Cohort 1 (C1A+C1B), PBTZ169 | Cohort 2 (C2), PBTZ169 | Cohort 3 (C3), PBTZ169 | Cohort 4 (C4), PBTZ169 | Cohort 5 (C5), PBTZ169
Number analyzed (Participants) | 20 | 10 | 10 | 10 | 10
AEs
  Number of AEs | 9 | 4 | 5 | 2 | 9
  Number of SAEs | 0 | 0 | 0 | 0 | 0
  Number of drug-related AEs | 9 | 4 | 5 | 1 | 6
  Drug-related "Cardiac disorders" AEs | 3 | 0 | 1 | 0 | 0
  Drug-related "GastroInt." AEs | 1 | 1 | 1 | 1 | 2
  Drug-related "Investigations" AEs | 4 | 0 | 2 | 0 | 0
  Drug-related "Nervous syst." AEs | 1 | 3 | 1 | 0 | 2
  Drug-related "Metabolic" AEs | 0 | 0 | 0 | 0 | 2

2. Primary Outcome: Number of Subjects With AEs
Description: Safety and tolerability: number of subjects with adverse events
Time Frame: Up to last visit time point: C2, C3, C4 up to Day 7; C1 up to Day 13; C5 up to Day 21 after first drug intake
Population: Safety population
Measure: Number; unit: participants
Arm/Group | Cohort 1 (C1A+C1B), PBTZ169 | Cohort 2 (C2), PBTZ169 | Cohort 3 (C3), PBTZ169 | Cohort 4 (C4), PBTZ169 | Cohort 5 (C5), PBTZ169
Number analyzed (Participants) | 20 | 10 | 10 | 10 | 10
participants
  Number of sbjs with AEs | 6 | 3 | 5 | 2 | 6
  Number of sbjs with drug-related AEs | 6 | 3 | 5 | 1 | 5

3. Secondary Outcome: CS Changes in Vital Signs
Description: Safety and tolerability:Clinically significant changes in vital signs (blood pressure, HR, body temperature, RR)
Time Frame: Up to last visit time point: C2, C3, C4 up to Day 7; C1 up to Day 13; C5 up to Day 21 after first drug intake
Population: Safety population
Measure: Number; unit: No of cases of CS changes in vital signs
Arm/Group | Cohort 1 (C1A), PBTZ169 | Cohort 1 (C1B), PBTZ169 | Cohort 2 (C2), PBTZ169 | Cohort 3 (C3), PBTZ169 | Cohort 4 (C4), PBTZ169 | Cohort 5 (C5), PBTZ169
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
No of cases of CS changes in vital signs
  CS Changes in blood pressure | 0 | 0 | 0 | 0 | 0 | 0
  CS changes in HH: Sinus tachycardia | 0 | 3 | 0 | 0 | 0 | 0
  CS Changes in Temperature | 0 | 0 | 0 | 0 | 0 | 0
  CS Changes in RR | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: ECG Results (Safety and Tolerability)
Description: Clinically significant abnormal deviations in ECG findings
Time Frame: Up to last visit time point: C2, C3, C4 up to Day 7; C1 up to Day 13; C5 up to Day 21 after first drug intake
Population: Safety population
Measure: Number; unit: participants
Arm/Group | Cohort 1 (C1A), PBTZ169 | Cohort 1 (C1B), PBTZ169 | Cohort 2 (C2), PBTZ169 | Cohort 3 (C3), PBTZ169 | Cohort 4 (C4), PBTZ169 | Cohort 5 (C5), PBTZ169
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
participants
  Electrocardiogram repolarisation abnormality | 1 | 0 | 0 | 1 | 0 | 0
  Sinus tachycardia | 0 | 1 | 0 | 0 | 0 | 0
  Electrocardiogram abnormal | 0 | 0 | 0 | 1 | 0 | 0
  Defect conduction intraventricular | 0 | 0 | 0 | 1 | 0 | 0

5. Secondary Outcome: Laboratory Examinations Results (Safety and Tolerability)
Description: Complete blood count, biochemical blood test, urine analysis
Time Frame: Up to last visit time point: C2, C3, C4 up to Day 7; C1 up to Day 13; C5 up to Day 21 after first drug intake
Measure: Number; unit: participants
Arm/Group | Cohort 1 (C1A), PBTZ169 | Cohort 1 (C1B), PBTZ169 | Cohort 2 (C2), PBTZ169 | Cohort 3 (C3), PBTZ169 | Cohort 4 (C4), PBTZ169 | Cohort 5 (C5), PBTZ169
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
participants
  CS Blood glucose increase | 1 | 2 | 0 | 0 | 0 | 0
  CS Hypercreatininaemia | 0 | 0 | 0 | 0 | 0 | 2
  CS Anaemia | 0 | 0 | 0 | 0 | 0 | 1
  CS Haemoglobin decreased | 0 | 0 | 0 | 0 | 0 | 1
  CS Thrombocytosis | 0 | 0 | 0 | 0 | 0 | 1

6. Secondary Outcome: Results of Physical Examination: CS Deviations
Description: Safety and tolerability: number of physical examinations with CS deviations in results
Time Frame: Up to last visit time point: C2, C3, C4 up to Day 7; C1 up to Day 13; C5 up to Day 21 after first drug intake
Population: Safety population
Measure: Number; unit: CS physical examination deviations
Arm/Group | Cohort 1 (C1A), PBTZ169 | Cohort 1 (C1B), PBTZ169 | Cohort 2 (C2), PBTZ169 | Cohort 3 (C3), PBTZ169 | Cohort 4 (C4), PBTZ169 | Cohort 5 (C5), PBTZ169
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
CS physical examination deviations | 0 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Peak Plasma Concentration (Сmax)
Description: Сmax of PBTZ169 at the timepoints:
  C1A, C1B, C2 and C4: point 0 (-5 min to -1 min), 0:30, 1:00, 1:30, 2:00, 3:00, 4:00, 6:00, 9:00, 12:00, 24:00, 48:00 and 72:00 (h:min).
  C3 (two administrations): point 0 (-5 min to -1 min), 0:30, 1:00, 1:30, 2:00, 3:00, 4:00, 6:00, 9:00, 12:00 (the point before the second administration from -5 min to -1 min), 12:30, 13:00, 13:30, 14:00, 15:00, 16:00, 18:00, 21:00, 24:00, 48:00 , 72:00 (h:min) after the first administration of the medicinal product.
  C5 (14 days of intake): 5 minutes before the administration (only until the first dose), 0 min and within 24 h after the administration of the 1st, 7th and last (14th) dose: 0:15, 0:30, 1:00, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 10:00, 12:00, 24:00 (h:min after the administration of a dose of the medicinal product); at 48 h and 72 h points after the last (14th) dose of PBTZ169
Time Frame: In the dosing interval (up to 72 hours after the last drug administration)
Population: C1-4 - Single or double dose administration, C5 - Multiple administration for 14 days
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/ml
Groups:
- Cohort 1 (C1A+C1B), PBTZ169, Fasted; Cohort 1 (C1A+C1B), PBTZ169, After Meal: PBTZ169 640 mg OD: Two administrations once a day with a wash-out period: food effect
- Cohort 5 (C5), PBTZ169: Multiple administration of PBTZ169: 1280 mg once a day after meal for 14 days
  PBTZ169 1280 mg MD: Once a day after meals, 14 doses
Arm/Group | Cohort 1 (C1A+C1B), PBTZ169, Fasted | Cohort 1 (C1A+C1B), PBTZ169, After Meal | Cohort 2 (C2), PBTZ169 | Cohort 3 (C3), PBTZ169 | Cohort 4 (C4), PBTZ169 | Cohort 5 (C5), PBTZ169
Number analyzed (Participants) | 20 | 20 | 10 | 10 | 10 | 10
ng/ml
  Before dosing | 0.250 (0) | 0.250 (0) | 0.250 (0) | 0.250 (0) | 0.250 (0) | 0.250 (0)
  0.25 h: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10
  0.25 h |  |  |  |  |  | 0.250 (0)
  0.5 h | 10.701 (236.6) | 0.399 (199.6) | 19.351 (228.4) | 26.048 (131.0) | 24.576 (76.6) | 1.183 (864.4)
  1 h | 43.131 (84.5) | 8.827 (415.1) | 45.729 (100.8) | 48.328 (46.8) | 74.711 (52.4) | 22.877 (3056.8)
  1.5 h | 40.998 (108.3) | 59.226 (150.6) | 48.390 (81.1) | 45.679 (43.9) | 54.949 (66.3) | 109.319 (203.7)
  2 h | 33.660 (118.4) | 95.641 (113.9) | 43.633 (145.2) | 23.782 (46.9) | 39.253 (73.4) | 162.170 (141.1)
  3 h | 19.435 (106.4) | 90.330 (84.9) | 22.159 (167.4) | 11.438 (60.2) | 23.571 (75.4) | 128.518 (95.0)
  4 h | 10.775 (96.4) | 88.719 (50.2) | 15.773 (184.0) | 6.593 (73.8) | 13.897 (79.0) | 110.614 (68.7)
  6 h | 4.195 (75.3) | 31.083 (46.8) | 5.884 (171.9) | 3.461 (51.7) | 5.771 (73.0) | 68.001 (127.0)
  8 h: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10
  8 h |  |  |  |  |  | 34.331 (149.2)
  9 h: number analyzed (Participants) | 20 | 20 | 10 | 10 | 10 | 0
  9 h | 1.827 (77.4) | 10.815 (71.3) | 2.672 (166.7) | 1.330 (39.1) | 2.880 (87.8) |
  10 h: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10
  10 h |  |  |  |  |  | 14.636 (93.8)
  12 h | 1.144 (59.1) | 4.621 (55.6) | 1.944 (125.3) | 0.859 (51.7) | 1.440 (50.7) | 8.917 (73.8)
  12.5 h: number analyzed (Participants) | 0 | 0 | 0 | 10 | 0 | 0
  12.5 h |  |  |  | 6.247 (270.1) |  |
  13 h: number analyzed (Participants) | 0 | 0 | 0 | 10 | 0 | 0
  13 h |  |  |  | 26.515 (152.4) |  |
  13.5 h: number analyzed (Participants) | 0 | 0 | 0 | 10 | 0 | 0
  13.5 h |  |  |  | 54.520 (65.7) |  |
  14 h: number analyzed (Participants) | 0 | 0 | 0 | 10 | 0 | 0
  14 h |  |  |  | 41.996 (61.7) |  |
  15 h: number analyzed (Participants) | 0 | 0 | 0 | 10 | 0 | 0
  15 h |  |  |  | 23.165 (64.4) |  |
  16 h: number analyzed (Participants) | 0 | 0 | 0 | 10 | 0 | 0
  16 h |  |  |  | 13.113 (88.3) |  |
  18 h: number analyzed (Participants) | 0 | 0 | 0 | 10 | 0 | 0
  18 h |  |  |  | 8.351 (127.2) |  |
  21 h: number analyzed (Participants) | 0 | 0 | 0 | 10 | 0 | 0
  21 h |  |  |  | 3.590 (139.2) |  |
  24 h | 0.456 (106.1) | 1.428 (42.2) | 0.731 (85.5) | 1.763 (75.1) | 0.591 (55.8) | 4.695 (128.9)
  48 h: number analyzed (Participants) | 20 | 20 | 10 | 10 | 10 | 0
  48 h | 0.250 (0) | 0.385 (62.2) | 0.288 (47.1) | 0.383 (65.9) | 0.269 (23.6) |
  72 h: number analyzed (Participants) | 20 | 20 | 10 | 10 | 10 | 0
  72 h | 0.250 (0) | 0.260 (18.3) | 0.250 (0) | 0.269 (23.3) | 0.250 (0) |
  Day 7, before dosing: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10
  Day 7, before dosing |  |  |  |  |  | 8.352 (102.5)
  Day 7, 0.25 h: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10
  Day 7, 0.25 h |  |  |  |  |  | 8.424 (68.8)
  Day 7, 0.5 h: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10
  Day 7, 0.5 h |  |  |  |  |  | 15.488 (86.8)
  Day 7, 1 h: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10
  Day 7, 1 h |  |  |  |  |  | 102.727 (146.9)
  Day 7, 1.5 h: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10
  Day 7, 1.5 h |  |  |  |  |  | 196.799 (124.0)
  Day 7, 2 h: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10
  Day 7, 2 h |  |  |  |  |  | 247.253 (90.7)
  Day 7, 3 h: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10
  Day 7, 3 h |  |  |  |  |  | 214.245 (53.4)
  Day 7, 4 h: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10
  Day 7, 4 h |  |  |  |  |  | 163.523 (36.5)
  Day 7, 6 h: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10
  Day 7, 6 h |  |  |  |  |  | 71.494 (75.1)
  Day 7, 8 h: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10
  Day 7, 8 h |  |  |  |  |  | 34.724 (60.1)
  Day 7, 10 h: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10
  Day 7, 10 h |  |  |  |  |  | 21.163 (62.3)
  Day 7, 12 h: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10
  Day 7, 12 h |  |  |  |  |  | 13.464 (54.6)
  Day 7, 24 h: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10
  Day 7, 24 h |  |  |  |  |  | 6.509 (51.5)
  Day 14, befor dosing: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10
  Day 14, befor dosing |  |  |  |  |  | 7.657 (48.2)
  Day 14, 0.25 h: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10
  Day 14, 0.25 h |  |  |  |  |  | 7.625 (50.6)
  Day 14, 0.5 h: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10
  Day 14, 0.5 h |  |  |  |  |  | 12.027 (47.3)
  Day 14, 1 h: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10
  Day 14, 1 h |  |  |  |  |  | 56.489 (185.3)
  Day 14, 1.5 h: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10
  Day 14, 1.5 h |  |  |  |  |  | 150.856 (123.3)
  Day 14, 2 h: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10
  Day 14, 2 h |  |  |  |  |  | 208.562 (56.0)
  Day 14, 3 h: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10
  Day 14, 3 h |  |  |  |  |  | 205.471 (69.6)
  Day 14, 4 h: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10
  Day 14, 4 h |  |  |  |  |  | 189.609 (39.2)
  Day 14, 6 h: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10
  Day 14, 6 h |  |  |  |  |  | 81.751 (55.6)
  Day 14, 8 h: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10
  Day 14, 8 h |  |  |  |  |  | 42.315 (67.0)
  Day 14, 10 h: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10
  Day 14, 10 h |  |  |  |  |  | 28.824 (121.6)
  Day 14, 12 h: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10
  Day 14, 12 h |  |  |  |  |  | 14.270 (48.1)
  Day 14, 24 h: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10
  Day 14, 24 h |  |  |  |  |  | 6.040 (58.1)
  Day 14, 48 h: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10
  Day 14, 48 h |  |  |  |  |  | 2.128 (103.6)
  Day 14, 72 h: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10
  Day 14, 72 h |  |  |  |  |  | 0.360 (90.0)

8. Secondary Outcome: Trough Concentration With Repeated Administration (Ctrough)
Description: PBTZ169 concentration before drug intake (Days 2 - 15)
Time Frame: Up to 72 hours after the last drug administration
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/ml
Arm/Group | Cohort 5 (C5), PBTZ169
Number analyzed (Participants) | 10
ng/ml
  Day 2 | 4.695 (128.9)
  Day 3 | 4.502 (39.9)
  Day 4 | 6.243 (42.8)
  Day 5 | 6.874 (51.7)
  Day 6 | 6.585 (53.2)
  Day 7 | 8.352 (102.5)
  Day 8 | 6.509 (51.5)
  Day 9 | 7.422 (51.7)
  Day 10 | 6.664 (58.8)
  Day 11 | 6.433 (48.7)
  Day 12 | 6.006 (51.7)
  Day 13 | 5.942 (44.5)
  Day 14 | 7.657 (48.2)
  Day 15 | 6.040 (58.1)

9. Secondary Outcome: Time to Reach Maximum Concentration (Tmax)
Description: Cohort 3: Tmax relative to the time of administration in any dosage interval
Time Frame: Up to 72 hours after the last drug administration
Population: C1-4 - Single or double dose administration, C5 - Multiple administration for 14 days
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Cohort 1 (C1A+C1B), PBTZ169, Fasted | Cohort 1 (C1A+C1B), PBTZ169, After Meal | Cohort 2 (C2), PBTZ169 | Cohort 3 (C3), PBTZ169 | Cohort 4 (C4), PBTZ169 | Cohort 5 (C5), PBTZ169
Number analyzed (Participants) | 20 | 20 | 10 | 10 | 10 | 10
h
  Dosing day / Day 1 | 1.73 (0.896) | 2.90 (0.912) | 1.65 (0.709) | 1.35 (0.747) | 1.15 (0.242) | 2.60 (1.410)
  Day 7: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10
  Day 7 |  |  |  |  |  | 2.25 (0.825)
  Day 14: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10
  Day 14 |  |  |  |  |  | 2.40 (1.022)

10. Secondary Outcome: Plasma Half-life Time (T1/2)
Time Frame: Up to 72 hours after the last drug administration
Population: C1-4 - Single or double dose administration, C5 - Multiple administration for 14 days
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Cohort 1 (C1A+C1B), PBTZ169, Fasted | Cohort 1 (C1A+C1B), PBTZ169, After Meal | Cohort 2 (C2), PBTZ169 | Cohort 3 (C3), PBTZ169 | Cohort 4 (C4), PBTZ169 | Cohort 5 (C5), PBTZ169
Number analyzed (Participants) | 20 | 20 | 10 | 10 | 10 | 10
h
  Dosing day / Day 1 | 5.46 (3.134) | 7.68 (3.063) | 7.68 (2.043) | 6.33 (5.275) | 8.00 (4.258) | 10.07 (4.294)
  Day 7: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10
  Day 7 |  |  |  |  |  | 9.98 (3.357)
  Day 14: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10
  Day 14 |  |  |  |  |  | 14.81 (4.365)

11. Secondary Outcome: Area Under the Concentration-time Curve (AUC0 t)
Description: In the time interval from 0 to time (t) when the last blood sample is collected with a concentration above the limit of quantification.
  C5: for the data of Day 14 based on measurements within 72 hours after the last dose administration
Time Frame: Up to 72 hours after the last drug administration
Population: C1-4 - Single or double dose administration, C5 - Multiple administration for 14 days
Measure: Mean (Standard Deviation); unit: ng*h/ml
Arm/Group | Cohort 1 (C1A+C1B), PBTZ169, Fasted | Cohort 1 (C1A+C1B), PBTZ169, After Meal | Cohort 2 (C2), PBTZ169 | Cohort 3 (C3), PBTZ169 | Cohort 4 (C4), PBTZ169 | Cohort 5 (C5), PBTZ169
Number analyzed (Participants) | 20 | 20 | 10 | 10 | 10 | 10
ng*h/ml
  Dosing day / Day 1: number analyzed (Participants) | 20 | 20 | 10 | 10 | 10 | 0
  Dosing day / Day 1 | 181.63 (112.236) | 575.19 (221.735) | 258.42 (174.149) | 342.03 (141.061) | 220.77 (124.754) |
  Day 14: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10
  Day 14 |  |  |  |  |  | 1479.76 (459.066)

12. Secondary Outcome: Area Under the Concentration-time Curve (AUC0-∞)
Description: In the time interval from 0 to infinity
Time Frame: Up to 72 hours after the last drug administration
Population: C1-4 - Single or double dose administration, C5 - Multiple administration for 14 days
Measure: Mean (Standard Deviation); unit: ng*h/ml
Arm/Group | Cohort 1 (C1A+C1B), PBTZ169, Fasted | Cohort 1 (C1A+C1B), PBTZ169, After Meal | Cohort 2 (C2), PBTZ169 | Cohort 3 (C3), PBTZ169 | Cohort 4 (C4), PBTZ169 | Cohort 5 (C5), PBTZ169
Number analyzed (Participants) | 20 | 20 | 10 | 10 | 10 | 10
ng*h/ml
  Dosing day / Day 1 | 175.98 (104.828) | 584.06 (221.531) | 267.94 (175.918) | 348.56 (141.198) | 228.93 (124.855) | 1153.89 (482.189)
  Day 7: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10
  Day 7 |  |  |  |  |  | 1479.16 (594.599)
  Day 14: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10
  Day 14 |  |  |  |  |  | 1501.97 (483.483)

13. Secondary Outcome: Area Under the Concentration-time Curve (AUC0-24)
Description: C5 (multiple administration once a day for 14 days): AUC0-24 was calculated based on measurements within 24 hours after PBTZ169 intake
Time Frame: In the dosing interval (up to 24 hours after drug administration)
Population: C5 (multiple administration for 14 days) - AUC0-τ within 72 hours after the last (14th) dose administration
Measure: Mean (Standard Deviation); unit: ng/ml*h
Arm/Group | Cohort 5 (C5), PBTZ169
Number analyzed (Participants) | 10
ng/ml*h
  Day 1 | 1111.90 (463.267)
  Day 7 | 1374.48 (575.119)
  Day 14 | 1363.85 (450.006)

14. Secondary Outcome: Total Clearance (Clt/F)
Time Frame: Up to 72 hours after the last drug administration
Population: C1-4 - Single or double dose administration, C5 - Multiple administration for 14 days
Measure: Mean (Standard Deviation); unit: l/h
Arm/Group | Cohort 1 (C1A+C1B), PBTZ169, Fasted | Cohort 1 (C1A+C1B), PBTZ169, After Meal | Cohort 2 (C2), PBTZ169 | Cohort 3 (C3), PBTZ169 | Cohort 4 (C4), PBTZ169 | Cohort 5 (C5), PBTZ169
Number analyzed (Participants) | 20 | 20 | 10 | 10 | 10 | 10
l/h
  Dosing day / Day 1 | 4910.09 (2711.818) | 1260.08 (491.974) | 8246.42 (12883.377) | 4185.23 (1507.230) | 6617.74 (2217.282) | 1302.31 (548.472)
  Day 7: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10
  Day 7 |  |  |  |  |  | 959.89 (269.654)
  Day 14: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10
  Day 14 |  |  |  |  |  | 924.97 (261.681)

15. Secondary Outcome: Volume of Distribution (Vd/F)
Time Frame: Up to 72 hours after the last drug administration
Population: C1-4 - Single or double dose administration, C5 - Multiple administration for 14 days
Measure: Mean (Standard Deviation); unit: l
Arm/Group | Cohort 1 (C1A+C1B), PBTZ169, Fasted | Cohort 1 (C1A+C1B), PBTZ169, After Meal | Cohort 2 (C2), PBTZ169 | Cohort 3 (C3), PBTZ169 | Cohort 4 (C4), PBTZ169 | Cohort 5 (C5), PBTZ169
Number analyzed (Participants) | 20 | 20 | 10 | 10 | 10 | 10
l
  Dosing day / Day 1 | 33460.07 (19725.828) | 13475.58 (6895.800) | 67278.30 (61222.530) | 34649.86 (29430.057) | 77814.43 (50236.867) | 21126.27 (15900.286)
  Day 7: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10
  Day 7 |  |  |  |  |  | 13745.97 (5520.697)
  Day 14: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10
  Day 14 |  |  |  |  |  | 19411.17 (6813.126)

16. Secondary Outcome: Elimination Constant Kel
Time Frame: Up to 72 hours after the last drug administration
Population: C1-4 - Single or double dose administration, C5 - Multiple administration for 14 days
Measure: Mean (Standard Deviation); unit: 1/h
Arm/Group | Cohort 1 (C1A+C1B), PBTZ169, Fasted | Cohort 1 (C1A+C1B), PBTZ169, After Meal | Cohort 2 (C2), PBTZ169 | Cohort 3 (C3), PBTZ169 | Cohort 4 (C4), PBTZ169 | Cohort 5 (C5), PBTZ169
Number analyzed (Participants) | 20 | 20 | 10 | 10 | 10 | 10
1/h
  Dosing day / Day 1 | 0.1765 (0.1067) | 0.1027 (0.0356) | 0.0993 (0.0396) | 0.1865 (0.1175) | 0.1154 (0.0682) | 0.0866 (0.0501)
  Day 7: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10
  Day 7 |  |  |  |  |  | 0.0765 (0.0240)
  Day 14: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10
  Day 14 |  |  |  |  |  | 0.0512 (0.0180)

17. Secondary Outcome: Relative Bioavailability
Description: f=AUC0-∞(T)/AUC0-∞(R); f'=AUC0-t(T)/AUC0-t(R) Test (T) - PBTZ169 640 mg after meals, reference (R) - PBTZ169 640 mg fasted
Time Frame: Up to 72 hours after the last drug administration
Measure: Geometric Mean (90% Confidence Interval); unit: % of T/R geometric mean ratio
Groups:
- Cohort 1 (C1A+C1B), PBTZ169, "After Meals (T)"/"Fasted (R)": PBTZ169 640 mg OD: Two administrations once a day with a wash-out period (cross-over): food effect
Arm/Group | Cohort 1 (C1A+C1B), PBTZ169, "After Meals (T)"/"Fasted (R)"
Number analyzed (Participants) | 20
% of T/R geometric mean ratio
  f | 344.54 [293.99 to 403.80]
  f' | 350.20 [300.94 to 407.52]

18. Secondary Outcome: Relative Degree of Absorption
Description: f"=Cmax(T)/Cmax(R). Test (T) - PBTZ169 640 mg after meals, reference (R) - PBTZ169 640 mg fasted
Time Frame: Up to 72 hours after the last drug administration
Measure: Geometric Mean (90% Confidence Interval); unit: geometric mean ratio, %
Arm/Group | Cohort 1 (C1A+C1B), PBTZ169, "After Meals (T)"/"Fasted (R)"
Number analyzed (Participants) | 20
geometric mean ratio, % | 229.03 [179.29 to 292.56]

19. Secondary Outcome: Number of Subjects With CS Changes in Vital Signs
Description: Safety and tolerability: No. of sbjs with clinically significant changes in vital signs (blood pressure, HR, body temperature, RR)
Time Frame: Up to last visit time point: C2, C3, C4 up to Day 7; C1 up to Day 13; C5 up to Day 21 after first drug intake
Population: Safety population
Measure: Number; unit: participants
Arm/Group | Cohort 1 (C1A), PBTZ169 | Cohort 1 (C1B), PBTZ169 | Cohort 2 (C2), PBTZ169 | Cohort 3 (C3), PBTZ169 | Cohort 4 (C4), PBTZ169 | Cohort 5 (C5), PBTZ169
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
participants
  CS Blood pressure deviations | 0 | 0 | 0 | 0 | 0 | 0
  CS Sinus tachycardia | 0 | 1 | 0 | 0 | 0 | 0
  CS Temperature changes | 0 | 0 | 0 | 0 | 0 | 0
  CS RR changes | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Single and double dosing groups - up to 5 ± 1 days after the last PBTZ169 dose intake (Cohorts 1-4): C1A, C1B - up to Day 12 ± 1 (Day 1 - 1st dosing day) C2, C3, C4 - up to Day 6 ± 1 (Day 1 - dosing day) Multiple dosing group - up to 7 ± 1 days after the last PBTZ169 dose intake (Cohort 5): C5 - up to Day 21±1 (Day 1 - 1st dosing day)
Arm/Group | Cohort 1 (C1A+C1B), PBTZ169 | Cohort 2 (C2), PBTZ169 | Cohort 3 (C3), PBTZ169 | Cohort 4 (C4), PBTZ169 | Cohort 5 (C5), PBTZ169
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/10 | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/10 | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 6/20 | 3/10 | 5/10 | 1/10 | 5/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (C1A+C1B), PBTZ169 (N=20) | Cohort 2 (C2), PBTZ169 (N=10) | Cohort 3 (C3), PBTZ169 (N=10) | Cohort 4 (C4), PBTZ169 (N=10) | Cohort 5 (C5), PBTZ169 (N=10)
Sinus tachycardia (Cardiac disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Defect conduction intraventricular (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram abnormal (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram repolarisation abnormality (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 1 (2)
Hypercreatininaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-11): https://cdn.clinicaltrials.gov/large-docs/24/NCT04150224/Prot_SAP_000.pdf